CLINICAL TRIAL: NCT02931240
Title: Clinical Study of the BioVentrix Revivent TC™ System for Treatment of Left Ventricular Aneurysms (ALIVE)
Brief Title: BioVentrix Revivent TC™ System Clinical Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BioVentrix (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIP-0066
Record Dates: First submitted 2016-09-30; First posted 2016-10-13 (Estimated); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Ventricular Dysfunction, Left
MeSH Terms: conditions — Ventricular Dysfunction, Left

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Treatment (Experimental): Treatment with the Revivent TC System
  Interventions: Device: Revivent TC
- Control Pool (No Intervention): Treatment with Guideline Directed Medical Therapy for Heart Failure Symptoms Only

INTERVENTIONS:
Device: Revivent TC — Treatment of LV scar
  Arms: Treatment

SUMMARY:
A prospective, multi-center, dual-arm pivotal study of the BioVentrix Revivent TC System, with 2:1 study vs. active concurrent control group allocation ratio. This study will include 126 patients of which 84 patients will be treated with the investigational device and 42 patients will be included in an active control group.

DETAILED DESCRIPTION:
The Revivent TC System is indicated for patients referred for surgical treatment of left ventricular scar that is contiguous, and includes both anterior and septal components. Primary and Secondary Effectiveness Endpoints will compare data from the patients treated with the Revivent TC System to a control pool of patients who comply with all aspects of the protocol except scar location and are not treated with the investigational devices but remain on Guideline Directed Medical Therapy (GDMT). The primary safety and effectiveness endpoints will be evaluated at 12 months post procedure. The study will be conducted at a maximum of 20 clinical centers.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* LV Aneurysm or Scar Presence: Defined by presence of a contiguous acontractile (akinetic and/or dyskinetic) scar;
* LV Aneurysm/Scar Location: Defined as a scar involving septum and/or anterior, apical or anterolateral regions of the left ventricle as evidenced by cardiac imaging and referred for surgical management;
* Viability of myocardium in regions remote from area of intended scar exclusion as evidenced by cardiac imaging;
* Left Ventricular Ejection Fraction < 45%;
* Left ventricular end-systolic volume index ≥50 mL/m2;
* Suffering from heart failure symptoms as defined by NYHA Classification > 2 not responsive to medical therapy;
* Patient completed 6 Minute Walk Test and MLHF Quality of Life Questionnaire (can be performed at baseline visit);
* Patient is on adequate Guideline Directed Medical Therapy (GDMT);
* Subject or a legally authorized representative must provide written informed consent;
* Agree to required follow-up visits; and
* Female subject of childbearing potential does not plan pregnancy for at least one year following the index procedure. For a female of childbearing potential, a pregnancy test must be performed with negative results known within seven days prior to index procedure Candidates for the study group must meet ALL of the inclusion criteria.

Candidates allocated to active concurrent control pool of patients must meet all inclusion criteria (including LV Aneurysm/Scar Presence), WITH THE EXCEPTION OF ONE OF THE FOLLOWING:

* They have undergone previous pericardiotomy, left thoracotomy, or open heart surgery, or
* The LV Aneurysm/Scar location does not permit treatment with the study device, or
* The patient elects to be enrolled in the control group

Exclusion Criteria:

Candidates will be excluded from the study and active concurrent control group if ANY of the following conditions are present:

* Cardiac Resynchronization Therapy (CRT) or ICD pacing lead placement ≤ 60 days prior to enrollment;
* Valvular heart disease, which in the opinion of the investigator, will require surgery;
* Functional Mitral Regurgitation greater than moderate (i.e. EROA>20mm sq.) and degenerative MR (including MR due to papillary muscle rupture);
* Need for coronary revascularization, in the opinion of the site investigator;
* Peak Systolic Pulmonary Arterial Pressure > 60 mm Hg via echo or right heart catheterization and/or evidence of cor pulmonale;
* Myocardial Infarction within 90 days prior to enrollment;
* Within the last six months, a prior CVA or TIA, or any intracranial hemorrhage, or any permanent neurologic deficit, or any known intracranial pathology;
* Co-morbid disease process with life expectancy of less than one year or active malignancy not in remission;
* Any solid organ transplant or is on waiting list for any solid organ transplant other than cardiac;
* Chronic renal failure with a serum creatinine >2.5 mg/dL and/or GFR<30ml/min;
* Subject is currently participating in another clinical trial that has not yet completed its primary endpoint;
* Presence of significant ventricular arrhythmias

The following exclusion criteria apply only to the treatment group and do not apply to the concurrent control cohort:

* Contraindication or inability to adhere to systemic anticoagulation;
* Known hypersensitivity or contraindication to device materials;
* Previous pericardiotomy or left thoracotomy;
* Pathology/previous surgery/radiation therapy of the right neck that would interfere with placement of a 14F delivery catheter;
* Prior open heart surgery or significant pericarditis;
* Calcified ventricular wall in the area of intended anchor implants as verified by cardiac imaging;
* Thrombus or intra-ventricular mass in the left atrium or ventricle as verified by cardiac imaging that has not been adequately treated with anticoagulant.
* Functioning pacemaker leads in antero-apical RV, which, in the opinion of the investigator, would interfere with anchor placement;

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2017-08-29 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of all cause death, mechanical support, emergent cardiac surgery, prolonged mechanical ventilation, renal failure and clinically important stroke compared to data from the STS database for surgical LV aneurysm repair. | 1 Month
  Composite primary safety endpoint of all cause death, placement of a mechanical support device intra or post-op (IABP, VAD, ECMO or catheter based), emergent cardiac surgery including reoperation for bleeding or tamponade, prolonged mechanical ventilation, renal failure and clinically important stroke (Rankin Score of 4 or higher) through 30-days post procedure. Data from the patients treated with the Revivent TC System will be compared to surgical outcomes data from the Society for Thoracic Surgery database for surgical LV aneurysm repair.
The rate of all cause of death, mechanical support, and operation (or re-operation) for HF, bleeding or tamponade from 1 through 12 months post procedure compared to untreated patients who remain on Guideline Directed Medical Therapy (GDMT). | 1 Year
  A composite of all cause of death, placement of a mechanical support device and operation (or re-operation) for HF, bleeding or tamponade from 1 through 12 months (day 31 through 365) post procedure. Data from patients treated with the Revivent TC System will be compared to data from a control pool of patients who comply with all aspects of the protocol except scar (aneurysm) location and are not treated with the investigational devices remain on Guideline Directed Medical Therapy (GDMT). Patients in the GDMT group will be evaluated from day 31 through 365 after the date of enrollment into the study.

SECONDARY OUTCOMES:
The rate of re-hospitalization and improvement of HF Symptoms in patients treated with the test device compared to patients who are maintained on Guideline Directed Medical Therapy. | 1 year
  Composite primary effectiveness endpoint consisting of:
  * No hospital readmission for new or worsening heart failure, and
  * Improvement in MLHF Quality of Life score by >10 points, and
  * Improvement in 6 Minute Walk Distance by >25 meters, and
  * Improvement in NYHA Classification > 1 grade.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew S Wechsler, MD, Principal Investigator — Drexel University College of Medicine; Gregg W Stone, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai; Jerry D Estep, MD, Principal Investigator — The Cleveland Clinic
Locations (30):
- United States (25):
  - University of Arizona College of Medicine - Phoenix Banner University Medicine Heart Institute, Phoenix, Arizona
  - Ronald Regan UCLA Medical Center, Los Angeles, California
  - University of California, San Francisco, San Francisco, California
  - Los Robles Hospital & Medical Center, Thousand Oaks, California
  - Baptist Hospital of Maimi, Miami, Florida
  - Emory University Hospital Midtown, Atlanta, Georgia
  - WellStar Health System, Marietta, Georgia
  - Memorial Medical Center, Springfield, Illinois
  - Terrebonne General Medical Center, Houma, Louisiana
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Mount Sinai Hospital, New York, New York
  - New York Presbyterian Hospital, New York, New York
  - Wake Forest Baptist Hospital, Winston-Salem, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - UPMC Pinnacle, Harrisburg, Pennsylvania
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - CHI St. Luke's Health-Baylor St. Luke's Medical Center, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Winchester Medical Center, Winchester, Virginia
- Nemocnice Na Homolce, Prague, Czechia
- Greece (2):
  - Hygeia Hospital, Athens
  - Interbalkan Medical Center, Thessaloniki
- United Kingdom (2):
  - Papworth Hospital NHS Foundation Trust, Cambridge
  - Freeman Hospital, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Estep JD, Ben-Yehuda O, Wechsler AS, Puri R, Kao AC, Heimes JK, Pfeiffer MP, Boehmer JP, Ninios V, Zaman A, Stone GW. Transcatheter Left Ventricular Reconstruction in Heart Failure Patients With Prior Anterior Myocardial Infarction: The Prospective ALIVE Trial. JACC Heart Fail. 2025 Feb;13(2):296-308. doi: 10.1016/j.jchf.2024.09.023. Epub 2025 Jan 8. PMID 39797846
- See also: Sponsor Web Site — http://www.bioventrix.com